CLINICAL TRIAL: NCT01638390
Title: Use of the VisuMax™ Femtosecond Laser Lenticule Removal Procedure for the Correction of Myopia
Brief Title: Use of the VisuMax™ Femtosecond Laser
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Carl Zeiss Meditec, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VISUMAX-2012-1
Record Dates: First submitted 2012-07-02; First posted 2012-07-11 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2018-12

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment of Myopia (Other): The reduction or elimination of myopia from ≥ -1.00 D to ≤ -8.00 D with ≤ -0.50 D cylinder and MRSE ≤ -8.25 D.
  Interventions: Device: Treatment with the VisuMax™ Femtosecond Laser

INTERVENTIONS:
Device: Treatment with the VisuMax™ Femtosecond Laser — The reduction or elimination of myopia from ≥ -1.00 D to ≤ -8.00 D with ≤ -0.50 D cylinder and MRSE ≤ -8.25 D.
  Other Names: VisuMaxTM Femtosecond Laser

SUMMARY:
The objective of this clinical trial is to evaluate the safety and effectiveness of the Carl Zeiss Meditec VisuMax™ Femtosecond Laser lenticule removal procedure for the reduction or elimination of myopia from ≥ -1.00 D to ≤ -8.00 D with ≤ -0.50 D cylinder and MRSE (Manifest Refractive Spherical Equivalent) ≤ -8.25 D.

DETAILED DESCRIPTION:
This is a prospective multi-center clinical trial in which a total of 360 eyes of consecutive subjects will be enrolled, treated with the VisuMax™ Femtosecond Laser, and followed for a 12-month period. The study will be conducted at up to 8 clinical sites.

Enrollment will be phased such that 100 eyes will be initially enrolled and followed. When 50 of the initial eyes have reached the 3-month follow-up exam, an interim clinical study report will be submitted to FDA along with a request to continue enrollment up to 360 eyes.

Subjects will be screened for eligibility, and informed consent will be obtained from those who meet screening criteria and are interested in participating in the study. Eligible subjects will be examined preoperatively to obtain a medical history and to establish a baseline ocular condition. Baseline and postoperative measurements will include manifest refraction, cycloplegic refraction, distance visual acuity (best corrected and uncorrected), slit-lamp examination, fundus examination, corneal topography, central corneal pachymetry, mesopic pupil measurement, wavefront analysis, mesopic contrast sensitivity, and intraocular pressure (IOP).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects age 22 years of age and older;
* Spherical myopia from ≥ -1.00 D to ≤ -8.00 D, with ≤ -0.50 D cylinder and MRSE ≤ -8.25 D in the eye to be treated;
* A stable refraction for the past year, as demonstrated by a change in MRSE of ≤ 0.50 D in the eye to be treated;
* A difference between cycloplegic and manifest refractions of < 0.75 D spherical equivalent in the eye to be treated;
* UCVA worse than 20/40 in the eye to be treated;
* BSCVA at least 20/20 in the eye to be treated;
* Discontinue use of contact lenses for at least 2 weeks (for hard lenses) or 3 days (for soft lenses) prior to the preoperative examination, and through the day of surgery;
* All contact lens wearers must demonstrate a stable refraction (within ±0.5 D), as determined by MRSE, on two consecutive examinations at least 1 week apart, in the eye to be treated;
* Central corneal thickness of at least 500 microns in the eye to be treated;
* Willing and able to return for scheduled follow-up examinations;
* Able to provide written informed consent and follow study instructions in English.

Exclusion Criteria:

* Mesopic pupil diameter > 8.0 mm;
* Cylinder > -0.50 D;
* Treatment depth is less than 250 microns from the corneal endothelium;
* Eye to be treated is targeted for monovision;
* Fellow eye has BSCVA worse than 20/40;
* Abnormal corneal topographic findings, e.g. keratoconus, pellucid marginal degeneration in either eye;
* History of or current anterior segment pathology, including cataracts in the eye to be treated;
* Clinically significant dry eye syndrome unresolved by treatment in either eye;
* Residual, recurrent, active ocular or uncontrolled eyelid disease, corneal scars or other corneal abnormality such as recurrent corneal erosion or severe basement membrane disease in the eye to be treated;
* Ophthalmoscopic signs of progressive or unstable myopia or keratoconus (or keratoconus suspect) in either eye;
* Irregular or unstable (distorted/not clear) corneal mires on central keratometry images in either eye;
* History of ocular herpes zoster or herpes simplex keratitis;
* Deep orbits, strong blink, anxiety, pterygium, or any other finding suggesting difficulty in achieving or maintaining suction;
* Difficulty following directions or unable to fixate;
* Previous intraocular or corneal surgery of any kind in the eye to be treated, including any type of surgery for either refractive or therapeutic purposes;
* History of steroid-responsive rise in intraocular pressure, glaucoma, or preoperative IOP > 21 mmHg in either eye;
* History of diabetes, diagnosed autoimmune disease, connective tissue disease or clinically significant atopic syndrome;
* Immunocompromised or requires chronic systemic corticosteroids or other immunosuppressive therapy that may affect wound healing;
* History of known sensitivity to planned study medications;
* Participating in any other ophthalmic drug or device clinical trial during the time of this clinical investigation;
* Pregnant, lactating, or of child-bearing potential and not practicing a medically approved method of birth control.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2012-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Dishler, M.D., Principal Investigator — Dishler Laser Institute; John Doane, M.D., Principal Investigator — Discover Vision Centers; Vance Thompson, M.D., Principal Investigator — Vance Thompson Vision Clinic, Prof., LLC; William Culbertson, M.D., Principal Investigator — Bascom Palmer Eye Institute; Sonia Yoo, M.D., Principal Investigator — Bascom Palmer Eye Institute; John Vukich, M.D., Principal Investigator — Davis Duehr Dean
Locations (5):
- United States (5):
  - Dishler Laser Institute, Greenwood Village, Colorado
  - Bascom Palmer Eye Institute, Miami, Florida
  - Discover Vision Centers, Leawood, Kansas
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Davis Duehr Dean, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment of Myopia
Started | 357 (enrolled)
Completed | 336 (treated eyes)
Not Completed | 21
Not completed — screening failures | 21

BASELINE CHARACTERISTICS:
Arm/Group | Treatment of Myopia
Number analyzed (Participants) | 336
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.33 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196
  Male | 140
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 309
  black | 10
  asian | 6
  other | 11
Surgical Eye [Count of Participants; unit: Participants]
  right | 152
  left | 184

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness- Predictability
Description: Number of participants with a decrease in manifest refraction spherical equivalent (MRSE) to within ± 1.00 D and ± 0.50 D of the intended refractive outcome at the point at which stability is first reached. The MRSE is the amount of prescription needed to obtain your best corrected vision as compared to your preoperative best corrected vision. A minimum of 75% of eyes should have an achieved refraction within ± 1.00 D of the intended outcome, and at least 50% of eyes should be within ± 0.50 D of the intended outcome.
Time Frame: 12 months
Population: The number reflected at the 12 month visit is the effectiveness population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment of Myopia
Number analyzed (Participants) | 310
Participants
  MRSE, Attempted vs. Achieved, ±0.50 D | 291
  MRSE, Attempted vs. Achieved, ±1.00 D | 306

2. Primary Outcome: Effectiveness- Improvement in UCVA Following Treatment
Description: Number of participants with uncorrected visual acuity (UCVA) of 20/40 or better at the point of stability. .This is vision without any form of prescription. A target of 85% of participants is required.
Time Frame: 12 month
Population: The number reflected at the 12 month visit is the effectiveness population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment of Myopia
Number analyzed (Participants) | 310
Participants | 309

3. Primary Outcome: Stability Criteria- Change Between Visits Within 1.00 Diopter (D)
Description: Number of participants with a change in postoperative refraction within 1.00 D between the 3 and 6 month visits. Stability was identified at the 6 month visit for the study.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Treatment of Myopia: Participants within 1.00 D change
Arm/Group | Treatment of Myopia
Number analyzed (Participants) | 327
Participants | 327

4. Primary Outcome: Safety- Preservation of Best-Spectacle Corrected Visual Acuity (BSCVA)
Description: 1. Number of participants with worse than 20/40 visual acuity with a preoperative BSCVA (Best Spectacle Corrected Visual Acuity) 20/20 or better. Target is less than 1% of study participants.
  2. Less than 5% of participants with BCVA loss ≥ 2 lines
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment of Myopia
Number analyzed (Participants) | 336
Participants
  BSCVA worse than 20/40 if 20/20 or better preopera | 0
  Loss of ≥ 2 lines BSCVA | 0

5. Primary Outcome: Safety- Induced Manifest Refractive Astigmatism
Description: Number of participants with an increase of astigmatism of greater than 2.00 D cylinder from the preoperative values. Target is less than 5% of participants.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment of Myopia
Number analyzed (Participants) | 336
Participants | 0

6. Primary Outcome: Safety- Adverse Events
Description: Number of participants for each type of adverse event. Target of less than 1% of participants for each type of adverse event.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Treatment of Myopia: Reported Adverse Events
Arm/Group | Treatment of Myopia
Number analyzed (Participants) | 336
Participants
  Retinal vasculitis | 1
  Carcinoma in situ, conjunctival | 1
  Decrease in BSCVA of ≥ 2 lines (≥10 letters) not d | 1
  Conjunctivitis, allergic | 1
  Conjunctivitis, viral | 1
  Herpetic lid and corneal lesion | 1
  Iritis | 1
  posterior vitreous detachment | 1
  Pyogenic Granuloma | 1
  Retained tissue, small | 2
  Difficult lenticule removal with tissue damage | 2

7. Primary Outcome: Safety- Contrast Sensitivity
Description: Number of participants who increased, remained the same, and decreased in contrast sensitivity. There are 4 different frequencies (1.5, 3.0, 6.0, and 12.0) which will be tested and are more difficult to detect as the frequency number increases.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Treatment of Myopia: Change in contrast sensitivity
Arm/Group | Treatment of Myopia
Number analyzed (Participants) | 310
Participants
  Gained at greater than or equal to 2 frequencies | 72
  No change | 232
  Loss at greater than or equal to 2 frequencies | 5

8. Primary Outcome: Stability Criteria- Change Between Visits Within 0.50 Diopter (D)
Description: Number of participants with a change in postoperative refraction within 0.50 D between the 3 and 6 month visits. Stability was identified at the 6 month visit for the study.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Groups:
- Treatment of Myopia: Participants within 0.50 D change
Arm/Group | Treatment of Myopia
Number analyzed (Participants) | 327
Participants | 317

9. Secondary Outcome: Safety- Patient Symptoms
Description: A standardized quality of vision (QoV) questionnaire was used in the study. A score is generated and was used to compare the results from baseline to the 12 month visit. Number of participants who improved, stayed the same, or worsened with regards to the frequency, severity, and bothersomeness of symptoms are reported.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Treatment of Myopia: Quality of Vision Score Change from Preoperative
Arm/Group | Treatment of Myopia
Number analyzed (Participants) | 309
Participants
  Frequency: worse | 116
  Frequency: same | 71
  Frequency: improved | 122
  Severity: worse | 93
  Severity: same | 95
  Severity: improved | 121
  Bothersome: worse | 79
  Bothersome: same | 119
  Bothersome: improved | 111

ADVERSE EVENTS:
Time Frame: approximately 2 years, 11 months
Arm/Group | Treatment of Myopia
All-Cause Mortality (participants affected / at risk) | 0/336
Serious Adverse Events (participants affected / at risk) | 0/336
Other Adverse Events (participants affected / at risk) | 14/336
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment of Myopia (N=336)
Decrease in BSCVA of greater than or equal to 2 lines (Eye disorders) | 1 (1) — A decrease in best spectacle corrected visual acuity (BSCVA) of greater than or equal to 2 lines not due to irregular astigmatism as shown by hard contact lens refraction at 3 months or later
Viral conjunctivitis (Eye disorders) | 1 (1) — An inflammatory process of the conjunctiva due a virus.
Retinal vasculitis (Eye disorders) | 1 (1) — A retinal blood vessel inflammation seen inside the eye.
Conjunctival carcinoma in situ (Eye disorders) | 1 (1) — A cancerous growth on the conjunctiva.
Allergic conjunctivitis (Eye disorders) | 1 (1) — an inflammatory process of the conjunctiva due to an allergen.
Difficult lenticule removal with tissue damage (Eye disorders) | 2 (2) — During the surgical procedure, the process of removing the lenticule caused damage to the cornea around the incision site.
Herpetic lid and corneal lesion (Eye disorders) | 1 (1) — A lid lesion and a corneal finding associated with the herpes virus.
Iritis (Eye disorders) | 1 (1) — An inflammatory process of the iris.
Posterior vitreous detachment (Eye disorders) | 1 (1) — The gel within the eye starts to change consistency and starts to constrict within the eye.
Perforated cap (Eye disorders) | 1 (1) — During the surgical process, a hole was created in the corneal flap during the lenticule removal process.
Pyogenic granuloma (Eye disorders) | 1 (1) — A non-cancerous growth on the lower lid.
Retained tissue (Eye disorders) | 2 (2) — During the surgical process, a small amount of tissue was retained which was seen on observation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less